CLINICAL TRIAL: NCT06570967
Title: A Retrospective and Prospective Observational Study of Hyperthyroidism in Children
Brief Title: A Clinical Study of Hyperthyroidism in Children
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Shi Tang, Attending Physician, Shengjing Hospital
Other Study IDs: 1223
Record Dates: First submitted 2024-08-13; First posted 2024-08-26 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Methimazole(MMI) — The initial dose of methimazole was 0.2-0.8 mg/(kg▪d). This dose was subsequently reduced by 25% to 50% and adjusted to maintain euthyroidism, based on the results of serum thyroid hormone testing during follow-up.

SUMMARY:
This study intends to conduct a retrospective and prospective study on children with hyperthyroidism, and it is a non-intervention study to collect information on diagnosis and treatment and long-term follow-up of children with hyperthyroidism. To investigate the clinical characteristics, treatment effect, side effects and remission of hyperthyroidism in children, to analyze the predictive factors for the effect of antithyroid drug treatment, remission and recurrence after drug withdrawal, and to explore the risk factors related to the occurrence of antithyroid drug-related adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤14 years old
2. Initial diagnosis of hyperthyroidism

Exclusion Criteria:

1. Hyperthyroidism had been treated with medication in other hospitals,
2. History of autoimmune hepatitis, viral hepatitis, hematological diseases, bone marrow or liver transplantation,
3. Patients with incomplete clinical data

Ages: 29 Days to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population included male and female with hyperthyroidism aged no more than 14 years. Participants must have not been treated with medication in other hospitals, have no history of autoimmune hepatitis, viral hepatitis, hematological diseases, bone marrow or liver transplantation, and have complete clinical data.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Remission of hyperthyroidism in children treated with methimazole. Remission is defined as having clinical and biochemical euthyroidism(FT3, FT4 and TSH are normal) without methimazole treatment for at least 12 months. | 10 years
  To analyze the therapeutic effect of methimazole and the predictors of remission of hyperthyroidism after methimazole treatment.
Adverse effects of methimazole in the treatment of hyperthyroidism in children. Adverse effects are defined as having neutropenia (absolute neutrophil count< 1500/µL), liver dysfunction (AST or ALT> 60 IU/L), rash, arthralgia, myalgia, et al. | 1 year
  Analyze the adverse reaction of methimazole treatment in hyperthyroidism children. Explore the risk factors related to the occurrence of methimazole related adverse reactions.

SECONDARY OUTCOMES:
Relapse of hyperthyroidism in children treated with methimazole. Relapse was defined as having clinical and biochemical hyperthyroidism (FT3 and FT4 increased and TSH decreased) after discontinuation of methimazole. | 10 years
  The risk factors of relapse in children with hyperthyroidism treated with MMI were analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT06570967/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT06570967/ICF_001.pdf